CLINICAL TRIAL: NCT02624206
Title: Specificity of Flavor-Nutrient Learning: An fMRI Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-1669; P30DK056350 (NIH)
Record Dates: First submitted 2015-10-08; First posted 2015-12-08 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2015-11

CONDITIONS: Feeding Behavior; Inhibition (Psychology)
MeSH Terms: conditions — Feeding Behavior; Inhibition, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Juice A (Active Comparator): Half of the group to receive Juice A, a novel juice flavor.
  Interventions: Dietary Supplement: Juice A
- Juice B (Active Comparator): Half of the group to receive Juice B, a novel juice flavor different from Juice A.
  Interventions: Dietary Supplement: Juice B

INTERVENTIONS:
Dietary Supplement: Juice A — Subjects to be given juice daily for 3 weeks.
  Arms: Juice A
Dietary Supplement: Juice B — Subjects to be given juice daily for 3 weeks.
  Arms: Juice B

SUMMARY:
This is an etiology study designed to examine the how people's brains and behaviors respond to regularly consuming a beverage. Participants are assessed at 2 behavioral assessments (Wave 1 and Wave 2), 2 scans (at the BRIC), and at 9 'intervention' assessments (5-10mins) different time periods throughout the study. At their first assessment (W1) they are randomized into one of two juices.

DETAILED DESCRIPTION:
Study design and Participants The investigators randomly assigned participants to consume one of two novel flavored, high-sugar beverages daily for a 3-week period. The study included fMRI and behavioral assessments pre-/post-intervention and 9 study visits during the intervention period. 20, healthy-weight, young adults (10 female, 10 male; x̅ age = 23.3±3.4; x̅ BMI = 22.1±1.9; 5% Hispanic,10% Asian/Pacific Islanders, 85% European Americans) completed protocol seen in Figure 1a. Exclusion criteria were a body mass index (BMI; kg/m2) <18.5 or >26.5, sweetened (artificial or caloric) beverage consumption > 6 times/week, tobacco/e-cigarette use > 6 times/week, psychoactive medications or drugs more than > 1 time/month, pregnancy, head injury with a loss of consciousness, significant cognitive impairment, major medical problems, endorsement of disordered eating or current Axis I psychiatric disorder as assessed by online screener. Participants provided written informed consent; methods and procedures were approved by University of North Carolina at Chapel Hill's Institutional Review Board.

Intervention Interested participants completed a brief online screening survey those that appeared to qualify were scheduled for the baseline visit where inclusion and exclusion were confirmed and consent was reviewed and obtained. Participants were randomly assigned to one of the two juice conditions, stratified by sex. Once consented, participants completed the behavioral and perceptual measures at the baseline behavioral assessment. On a separate day participants completed the baseline neuroimaging assessment. The day following the neuroimaging assessment participants began the intervention period where they consumed their assigned juice daily for the 3-week period. During the intervention period participants came to our lab every Monday, Wednesday and Friday (9 total assessments) to: consume a portion of that day's juice in the lab, complete perceptual measures and a weight assessment, pick up the following day(s) juice, and return the empty bottles from the previous day(s). On Fridays, participants were given two bottles to consume and instructed to consume one per day and return the bottles on the following Monday. Empty bottles were returned to increase compliance. The follow-up neuroimaging assessment was scheduled such that participants completed the 3-week intervention, did not consume a juice for 24 hours and then were scanned. The follow-up behavioral assessment occurred within three days of the follow-up scan Figure 1b.

Beverages were selected to be: sweetened from sugar, i.e., not include high fructose corn syrup, and/or artificial sweeteners, have no artificial flavors, colors or preservatives, calorically equivalent to common sugar-sweetened beverages (e.g., soft drinks), be caffeine- and texture-free, and generally novel in flavor. The juices were eucaloric, had similar palatability, and easily distinguishable from one another. Prior to study initiation, pilot taste testing was completed in a small sample to insure both the novelty and equal palatability of the two juices to be included in the study. The resulting two beverages were: Apple-Cherry-Berry juice and Orange-Tangerine-Passionfruit juice. The 10 fl oz bottles of juice each contained 133 kcals, 31g of sugar. The juice logos were selected to be novel, of similar visual complexity, both in black and white, convey no information beyond a unique symbol, yet be easily distinguishable from one another. Each juice was presented in individual 10 fl oz bottles with the only identifier a sticker of the associated logo.

ELIGIBILITY:
Inclusion Criteria:

* BMIs between 19 and 25

Exclusion Criteria:

* Contraindicators of fMRI (e.g., metal implants, braces, or pregnancy)
* Symptoms of major psychiatric disorders (substance use disorders, conduct disorder, ADHD, major depression, bipolar disorder, anorexia nervosa, bulimia nervosa, binge eating disorder)
* Active weight loss dieting
* Use of psychoactive drugs (e.g., cocaine)
* Serious medical problems (e.g., diabetes)
* Smoking
* Dietary practices that do not allow intake of dairy products during the phone screen will be excluded

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Voxel-wise Blood Oxygen Level Dependent (BOLD) Using Functional Magnetic Resonance Imaging (fMRI) of Brain Activation Signals in Response to Beverage Taste and Logo: Percent Change in BOLD Activations Including Outliers | Baseline, Post-Intervention Assessment (about 3 weeks after baseline)
  The juice fMRI paradigm assessed evoked blood oxygen level dependent (BOLD) response to receipt of both juices and a tasteless solution, and logo-elicited anticipation of both juices and tasteless solution.
  The paradigm was controlled by in-house scripts written in MATLAB (Mathworks, Inc., Natick, MA). The visual stimuli were two juice logos, a tasteless logo, and a fixation cross. Each logo (4 seconds) signaled impending delivery of 0.5 mL of the associated juice/tasteless over 4 seconds, with the fixation cross otherwise presented. Participants were visually instructed on when to swallow. A jitter ranging from 5 to 13 (x̅ =8) seconds followed each trial. In total, the participants were presented 27 repeats of the events of interest over 3, 12 min runs.

SECONDARY OUTCOMES:
Change in Response Time to Logo as Measured in Behavioral Impulsivity Task | Baseline, Post-Intervention Assessment (about 3 weeks after baseline)
  The primary objective of the behavioral impulsivity task was to examine motor disinhibition as represented by response time to the beverage logos and control logos. Participants were instructed to respond as quickly and accurately as possible with a keyboard press when shown the target logo, but withhold their responses during presentation of other logos. Participants performed the task twice, each time depicting one of the beverage logos as the 'target' logo at both the pre- and post-intervention assessments. The order of which logo was the 'target' logo was in a counterbalanced. Each task consisted of 48 trials. Stimuli were presented and reaction times, commission and omission errors were recorded using the Presentation software package (Version 9, Neurobehavioral Systems, Davis, CA). Change in response time is calculated as a difference between baseline and post-intervention assessment average response time across 48 trials.
Change in Error Rate to Logo as Measured in Behavioral Impulsivity Task | Baseline, Post-Intervention Assessment (about 3 weeks after baseline)
  The secondary objective of the behavioral impulsivity task was to examine error rate in response to the beverage logos and control logos. Participants were instructed to respond as quickly and accurately as possible with a keyboard press when shown the target logo, but withhold their responses during presentation of other logos. Participants performed the task twice, each time depicting one of the beverage logos as the 'target' logo at both the pre- and post-intervention assessments. The order of which logo was the 'target' logo was in a counterbalanced. Each task consisted of 48 trials. Stimuli were presented and reaction times, commission and omission errors were recorded using the Presentation software package (Version 9, Neurobehavioral Systems, Davis, CA). Change in error rate is calculated as a difference between baseline and post-intervention assessment total number of commission and omission error across 48 trials.
Change score in Visual Analog Scale Ratings of Beverage Perceptual Measures | Baseline, Intervention Visits 1-9 (over 3 weeks), Post-Intervention Assessment (about 3 weeks after baseline)
  All visual analog scales were presented on a computer screen and completed one at a time. If the scale was assessing response to taste, the participant consumed a small amount of the beverage and completed the associated scales. Perceived pleasantness of, and desire to consume the two juices was measured using adapted labeled hedonic scales at pre-/post-intervention. Pleasantness was phrased 'How pleasant is this taste' and anchored by (-100) 'most unpleasant imaginable' to (100) 'most pleasant imaginable', and 'neutral' (0) in the middle. Desire followed a similar pattern using 'desire to consume' as the phrasing. Pleasantness and desire of the assigned juice was also evaluated at the 9 intervention assessments. Perceived hunger was assessed via cross-modal visual analog scales, anchored by (-100) 'I am not hungry at all' to (100) 'I have never been more hungry'. The change score was calculated from the slope of ratings plotted by time.
Change in Restrained Eating Subscale Score as measured on Dutch Eating Behavior Questionnaire. | Baseline, Post-Intervention Assessment (about 3 weeks after baseline)
  The Dutch Eating Behavior Questionnaire is a 33-item self-report measure designed to assess the type of eating behavior and is organized into 3 subscales (emotional eating, externally-induced eating, and restrained eating). Subjects rated the frequency of their eating behaviors using a 5-point scale, where 1=never, 2=seldom, 3=sometimes, 4=often, and 5=very often. The Restrained Eating subscale consisted of 10 items and the scores ranged from 10 (worse outcome) to 50 (better outcome). The change was calculated as the difference between scores at Baseline and Post-Intervention Assessment.
Changes in Food Pattern From Baseline to Post-Intervention Assessment by Food Frequency Questionnaire. | Baseline, Post-Intervention Assessment (about 3 weeks after baseline)
  The Food Frequency Questionnaire (FFQ) is a self-reported checklist of 76 foods and beverages with a frequency response section. Subjects report generally how often each item was consumed over a two-week period of time. The six possible responses are 1= never in the last two weeks, 2= 1-3 times in the last 2 weeks, 3= 4-6 times in the last 2 weeks, 4= 7-9 times in the last two weeks, 5= 10-13 times in the last 2 weeks, 6= daily or more in the last two weeks. Responses information is used to estimate daily caloric intake (number of kcal) and macronutrient content (percent calories from carbohydrate/fat/protein). Food pattern is assessed as an aggregate of these measures. Changes in food pattern will be assessed as a difference from baseline to post-intervention assessment.
Change in Food Craving as assessed by the Food Craving Inventory (FCI) Score Changes of Food Pattern From Baseline by Food Frequency Questionnaire During the Intervention | Baseline, Post-Intervention Assessment (about 3 weeks after baseline)
  The Food Craving Inventory is a 28-item instrument measuring the frequency over the past month of general cravings and cravings for specific types of foods, namely: high fats, sweets, carbohydrates/starches, and fast-food fats. Subjects rate how often they have experienced a craving for each food on a 5-point frequency scale, where 1=never, 2=rarely (once or twice), 3=sometimes, 4= often, 5= always/almost every day. Food craving score is calculated as a total sum, and the change score is calculated from the difference between baseline to post-intervention assessment.
Change in Hedonic Hunger as assessed by the Power of Food Scale (PFS) Score | Baseline, Post-Intervention Assessment (about 3 weeks after baseline)
  The Power of Food scale assesses reported appetitive drive, food reward responsivity, sensitivity to food cues in the environment, and the frequency of food-related thoughts. The 21-item scale prompts subjects to rate how much they agree with statements about hedonic hunger on a 5-point scale, where 1=do not agree at all, 2=agree a little, 3=agree somewhat, 4=agree, and 5=strongly agree. The change in total PFS score will be calculated from the difference between baseline to post-intervention assessment.
Change in Food Habits as assessed by the Yale Food Addiction Scale | Baseline, Post-Intervention Assessment (about 3 weeks after baseline)
  The Yale Food Addiction Scale (YFAS) was designed to identify participants who exhibit signs of possible food addiction to specific foods. The 9-item questionnaire is based on substance dependence criteria in the DSM-IV-TR, as well as on scales that have been used to assess behavioral addictions. Subjects rate how often they have experienced a possible food addictive behavior on a 5-point frequency scale, where 0=never, 1=once a month, 2=2-4 times per month, 3= 2-3 times per week, 4= 4+ times per week. The change in total score is calculated from the difference between baseline to post-intervention assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Burger, PhD, MPH, RD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Derived] Burger KS. Frontostriatal and behavioral adaptations to daily sugar-sweetened beverage intake: a randomized controlled trial. Am J Clin Nutr. 2017 Mar;105(3):555-563. doi: 10.3945/ajcn.116.140145. Epub 2017 Feb 8. PMID 28179221